CLINICAL TRIAL: NCT03029416
Title: A Randomized Phase 2 Study of Two Radiation Dose Schedules of Stereotactic Body Radiotherapy (SBRT) to Lung Metastases < 5cm in Dimension
Brief Title: Two Radiation Dose Schedules of SBRT to Lung Metastases < 5cm in Dimension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PRMC Administrative Disapproval - Slow accrual
Sponsor: Ronald McGarry (Other)
Responsible Party: Sponsor-Investigator, Ronald McGarry, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-MULTI-21; MCC-16-LUN-101 (Other: Univ of KY Markey Cancer Center)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Neoplasm Metastasis; Cancer; Radiation Therapy Complication
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: 30 Gy single fraction SBRT 18 Gy x three fractions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Fraction of SBRT (Experimental): Stereotactic Body Radiation Therapy delivered in a single session on one day
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Fractionated SBRT (Experimental): Stereotactic Body Radiation Therapy delivered in three to five fractions with one fraction delivered every other day
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Stereotactic Body Radiation Therapy using different fractionation schedules

SUMMARY:
30 Gy single fraction of SBRT for lung metastases will result in comparable oncologic outcomes to 18Gy in three fractions (or dosing to a BED </-100Gy at the discretion of the radiation oncologist) with respect to disease control and toxicity.

DETAILED DESCRIPTION:
Using two different doses of SBRT, this study will examine the 6-month local disease control rate (LDCR) of the SBRT-treated metastasis to determine the optimum dosing for SBRT in pulmonary metastases. This will allow us to establish baseline SBRT data, from which we will develop a second trial to examine sequencing of immunotherapy with SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of malignant carcinoma/sarcoma (any site) with metastasis to lung.
* Patients must not be eligible for therapy with curative intent (i.e. surgery, radiation, etc).
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* Age ≥18 years
* ECOG performance status >/= 2 (Karnofsky≥60%)).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with more than >/=3 metastatic lung lesions or any one lesion greater than 5 cm. and/or extensive metastatic disease outside the chest.
* Patients who are receiving any other investigational agents.
* Patients with active systemic, pulmonary, or pericardial infection.
* Pregnant or lactating women
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Chemotherapy concurrent with SBRT is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Local Disease Control Rates | 6 MONTHS
  Response defined by the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ronald McGarry, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No